CLINICAL TRIAL: NCT02513641
Title: Effect of 2-Week Nightly Moderate Hypoxia on Oral Glucose Tolerance in Individuals With Type 2 Diabetes
Brief Title: Effect of 2-Week Nightly Moderate Hypoxia on Glucose Tolerance in Individuals With Type 2 Diabetes
Acronym: SLEEPDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Eric Ravussin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 2015-018
Record Dates: First submitted 2015-07-28; First posted 2015-07-31 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moderate Hypoxia (Experimental): 2-weeks of nightly exposure (7-12 hrs per night) to moderate hypoxia (~2,400 meters) using the Hypoxico Altitude Training Systems device.
  Interventions: Device: Hypoxico Altitude Training Systems

INTERVENTIONS:
Device: Hypoxico Altitude Training Systems — Participants will sleep in a tent (which will fit his/her personal mattress) simulating an altitude of ~2,400 meters for 7-12 hours each night for a period of 14 days. Baseline testing measures will include a oral glucose tolerance test (OGTT) and body composition (iDXA). Post-treatment testing measures will include OGTT only.

SUMMARY:
The purpose of this study is to determine if 2 weeks of nightly exposure (7-12 hours per night) to moderate hypoxia (~2,400 meters or 7,500 feet) improves glucose metabolism in people with type 2 diabetes.

DETAILED DESCRIPTION:
Exposure to hypoxia has been advocated as a possible therapeutic aid against obesity. Indeed, our laboratory has provided the first evidence that intermittent, nightly exposure to moderate hypoxia is beneficial in improving insulin sensitivity in healthy obese patients and, therefore, lowers the risk of developing type 2 diabetes. Benefits included reduced fasting glucose levels and improved whole-body (skeletal muscle) and hepatic insulin sensitivity. Whether such intermittent hypoxia improves glucose metabolism in people with type 2 diabetes is unknown.

ELIGIBILITY:
INCLUSION CRITERIA:

* Aged 20-65 yrs
* Body mass index (BMI) < 55 kg/m2
* Body weight 450 lbs or less (to accommodate body composition assessment)
* Have either been diagnosed with type 2 diabetes, or fasting blood glucose between 125 and 200 mg/dL, or have a hemoglobin A1c ≥ 6.5%
* Non-smokers
* Weight stable over the previous 3 months (<3 kg fluctuation)
* Known diagnosis of sleep apnea and ownership of a continuous positive airway pressure (C-PAP) device that must be worn throughout the nights spent in the tent
* If no known presence of sleep apnea, be willing to spend one night in a sleep laboratory (Louisiana Sleep Foundation) to assess presence of sleep apnea

EXCLUSION CRITERIA:

* Diagnosed with T2DM ≥ 15 years ago
* Pregnant Women
* Current insulin treatment
* Treatment with sulfonylureas or glitinides
* Treatment with a GLP-1 agonist
* Any other diabetes medication other than an oral agent is exclusionary unless otherwise cleared by medical investigator.
* Chronic Obstructive Pulmonary Disease (COPD)
* Congestive heart failure
* Prior severe cardiovascular events such as stroke or myocardial infarction
* If treated for T2DM with other oral agent, no change in the treatment for 1 month before the study and the duration of the study
* Previously known diagnosis of sleep apnea without ownership of a continuous positive airway pressure (C-PAP) device or agreement to use owned CPAP device during the nights spent in the tent
* Presence of sleep apnea following a positive home sleep test (HST), or have unsafe oxyhemoglobin saturation levels (less than 78%) during a one night sleep monitoring assessment conducted at the Louisiana Sleep Foundation without ownership of a continuous positive airway pressure (C-PAP) device or agreement to use owned C-PAP device during the nights spent in the tent
* History of high altitude sickness
* History of altitude sickness
* Does not have access to a bed or sleeping surface equivalent to or smaller than a queen size mattress

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-12; Primary Completion 2018-04 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ravussin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate Hypoxia
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Moderate Hypoxia
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Weight, Continuous [Mean (Standard Deviation); unit: kg] | 117.8 (18.6)
Body mass index, Continuous [Mean (Standard Deviation); unit: kg/m^2] | 39.6 (5.8)
Percent body fat, Continuous [Mean (Standard Deviation); unit: percent] | 43 (8)
Fat mass, Continuous [Mean (Standard Deviation); unit: kg] | 50.5 (12.2)
Fat-free mass, Continuous [Mean (Standard Deviation); unit: kg] | 67.3 (14.0)
Systolic blood pressure, Continuous [Mean (Standard Deviation); unit: mmHg] | 121 (13)
Diastolic blood pressure, Continuous [Mean (Standard Deviation); unit: mmHg] | 74 (10)
Hemoglobin A1C, Continuous [Mean (Standard Deviation); unit: percent] | 6.8 (0.7)
Total cholesterol (TC), Continuous [Mean (Standard Deviation); unit: mg/dL] | 170 (36)
High-density lipoprotein cholesterol (HDL), Continuous [Mean (Standard Deviation); unit: mg/dL] | 55 (18)
Low-density lipoprotein cholesterol (LDL), Continuous [Mean (Standard Deviation); unit: mg/dL] | 95 (22)
Triglycerides, Continuous [Mean (Standard Deviation); unit: mg/dL] | 100 (39)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Insulin sensitivity was determined using an oral glucose tolerance test. Insulin sensitivity was estimated using the whole-body insulin sensitivity index (WBISI), also known as the Matsuda Index (unitless): WBISI = 10,000 / [square root of (Glu0 x Ins0) x (mean glucose x mean insulin during an oral glucose tolerance test)] where Glu0 and Ins0 denote baseline glucose and insulin concentrations.
Time Frame: Baseline and Post-Moderate Hypoxia (14 days)
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Moderate Hypoxia
Number analyzed (Participants) | 8
unitless
  Baseline Measure | 1.7 (0.7)
  Post-Moderate Hypoxia Measure | 2.2 (1.7)

2. Secondary Outcome: Insulin Secretion
Description: Insulin secretion was determined using an oral glucose tolerance test. Insulin secretion was estimated using the Insulinogenic Index (IGI), an index of first-phase insulin response, and calculated from the ratio of the increments of serum insulin to glucose measured at 30 minutes: IGI (unitless) = (Ins30 - Ins0)/(Glu30 - Glu0), where insulin and glucose from 0 and 30 minutes are used.
Time Frame: Baseline and Post-Moderate Hypoxia (14 days)
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Moderate Hypoxia
Number analyzed (Participants) | 8
unitless
  Baseline Measure | 0.6 (0.6)
  Post-Moderate Hypoxia Measure | 0.7 (0.7)

3. Secondary Outcome: Beta-cell Function
Description: Beta-cell function was determined using an oral glucose tolerance test. Beta-cell function was estimated by the Disposition Index, or the product of insulin sensitivity and insulin secretion: DI (unitless) = Matsuda Index (WBISI) x Insulinogenic Index (IGI).
Time Frame: Baseline and Post-Moderate Hypoxia (14 days)
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Moderate Hypoxia
Number analyzed (Participants) | 8
unitless
  Baseline Measure | 0.9 (1.0)
  Post-Moderate Hypoxia Measure | 1.4 (1.7)

4. Secondary Outcome: 2-hour Glucose Area-under-the-curve
Description: 2-hour glucose area-under-the-curve (mg/dL x hour) was determined using an oral glucose tolerance test.
Time Frame: 0, 0.5, 1, 1.5, and 2 hours at Baseline and Post-Moderate Hypoxia (14 days)
Measure: Mean (Standard Deviation); unit: mg/dL x hour
Arm/Group | Moderate Hypoxia
Number analyzed (Participants) | 8
mg/dL x hour
  Baseline Measure | 501 (99)
  Post-Moderate Hypoxia Measure | 439 (65)

5. Secondary Outcome: 2-hour Insulin Area-under-the-curve Via Oral Glucose Tolerance Test
Description: 2-hour insulin area-under-the-curve (μU/mL x hr) was determined using an oral glucose tolerance test.
Time Frame: 0, 0.5, 1, 1.5, and 2 hours at Baseline and Post-Moderate Hypoxia (14 days)
Measure: Mean (Standard Deviation); unit: uU/mL x hour
Arm/Group | Moderate Hypoxia
Number analyzed (Participants) | 8
uU/mL x hour
  Baseline Measure | 180 (154)
  Post-Moderate Hypoxia Measure | 168 (176)

ADVERSE EVENTS:
Time Frame: Approximately 1-month (baseline screening to end of 2-week moderate hypoxia exposure)
Arm/Group | Moderate Hypoxia
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Hypoxia (N=8)
Feelings of depression (Psychiatric disorders) | 1 (1)
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT02513641/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT02513641/ICF_001.pdf